CLINICAL TRIAL: NCT02639962
Title: Characteristics of Culprit Lesion and Changes in Plaque Composition During Follow up in NSTEMI. A Dual Energy Cardiac CT Study
Brief Title: Characteristics of Culprit Lesion and Changes in Plaque Composition. A Dual Energy Cardiac CT Study
Acronym: S-20130009
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Hussam Mahmoud Sheta, MD, Odense University Hospital
Other Study IDs: Challenge
Record Dates: First submitted 2015-12-09; First posted 2015-12-28 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Coronary Arteriosclerosis
Keywords: culprit lesion; arteriosclerosis; cardiac CT
MeSH Terms: conditions — Coronary Artery Disease; Arteriosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for analyses as hs-CRP, Interleukins and other inflammatory agents.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NSTEMI: patients hospitalized with NSTEMI diagnosed according to the national Danish guidelines, and are scheduled to coronary angiography.
  Interventions: Radiation: Cardiac CT
- patients with stable angina pectoris: Patients in this group have stable angina symptoms and had verified plaques by earlier CAG or Cardiac CT
  Interventions: Radiation: Cardiac CT

INTERVENTIONS:
Radiation: Cardiac CT — Cardiac CT before the CAG, and follow up after 2 month and 12 month

SUMMARY:
Identifying patients who are at risk for a future myocardial infarction, is still one of the biggest challenges in cardiology.

In this study the investigators will investigate culprit lesion in patients with NSTEMI and the ability of cardiac CT with dual energy computed tomography (DECT) scanning to describe and identify plaques that may be vulnerable. The investigators will also describe changes in characteristic in both stable and unstable plaques during 1 year follow up of NSTEMI and a matching group of stable angina pectoris (SAP) patients.

DETAILED DESCRIPTION:
Patients with verified NSTEMI undergo contrast-enhanced coronary DECT before conventional coronary angiography (CAG), and DECT characteristics of the culprit lesion will be determined. All Non-culprit lesions will be observed during 2 month and 1 year follow up characteristics and changes in plaque composition, volume and core content will be assessed.

Patients with SAP undergo a baseline DECT similar to NSTEMI group. Because the expected change in coronary plaques in SAP group is minimal, there is no need for follow up at 2 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSTEMI and scheduled to CAG or patients with SAP

Exclusion Criteria:

* Not suitable to undergo CT with contrast agent:
* Known allergy-like reactions to contrast or Claustrophobia
* Atrial fibrillation or significant arrhythmia judged to potentially limit quality of CT
* Known renal failure/insufficiency or s-creatinin> 140 µmol/L.
* Severe/symptomatic thyrotoxicosis
* pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with verified NSTEMI and Patients with SAP
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Description and characteristics of culprit lesion by DECT. (z-value) | 72 hours
  measure the z-value for the culprit lesion, by marking the culprit lesion with a region of interest (ROI) and the DECT will calculate the mean z-value by mg/mm^3 in the marked ROI

SECONDARY OUTCOMES:
Describe if the culprit lesion contains 1: soft 2: mixed or 3: calcified tissue | 72 hours
  Visually description if the culprit lesion contain
  1: soft tissue (dark area in the scan) 3: calc (white area) or 2: mixed (combined dark and white areas)
Measure the volume of the culprit lesion | 72 hours
  CT software will be automatically able to measure the volume (mm3) og culprit lesion
Measure the remodeling index of culprit lesion | 72 hours
  CT software will be automatically able to measure the remodeling index in culprit lesion (mm)
Determine the mean Z value for non-culprit plaques containing 1: soft tissue | 72 hours
  measure the z-value for the culprit lesion, by marking the lesion with a ROI and the DECT will calculate the mean z-value in the marked ROI
Determine the mean Z value for non-culprit plaques containing 1: soft tissue | 2 month
  measure the z-value for the culprit lesion, by marking the lesion with a ROI and the DECT will calculate the mean z-value mg/mm^3 in the marked ROI
Determine the mean Z value for non-culprit plaques containing 1: soft tissue | 1 year
  measure the z-value for the culprit lesion, by marking the lesion with a ROI and the DECT will calculate the mean z-value mg/mm^3 in the marked ROI
Determine the mean Z value for non-culprit plaques containing 2: mixed tissue | 72 hours
  z-value mg/mm^3
Determine the mean Z value for non-culprit plaques containing 2: mixed tissue | 2 month
  z-value mg/mm^3
Determine the mean Z value for non-culprit plaques containing 2: mixed tissue | 1 year
  z-value mg/mm^3
Determine the mean Z value for non-culprit plaques containing 3: calcified tissue | 72 hours
  z-value mg/mm^3
Determine the mean Z value for non-culprit plaques containing 3: calcified tissue | 2 month
  z-value mg/mm^3
Determine the mean Z value for non-culprit plaques containing 3: calcified tissue | 1 year
  z-value mg/mm^3
changes in non-culprit plaques during 1 year in comparison til patients with stable angina pectoris | 1 year
  z-value z-value mg/mm^3
z value in myocardium related to culprit vessel compared to z-value in myocardium corresponded to non-culprit vessel | 72 hours
  z-value z-value mg/mm^3

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, Study Director — Odense University Hospital, Svendborg Research Department
Locations (1):
- Department of Medical Research, OUH, Svendborg, Svendborg, Denmark